CLINICAL TRIAL: NCT05671003
Title: The Effect of Dentition, Eating Rate, Oral Processing, and Gastric Emptying on Appetite and Satiety in Older Adults (≥65 Years of Age)
Brief Title: Oral Processing and Appetite in Older Adults
Status: Completed | Type: Observational
Sponsor: University of Reading (Other)
Collaborators: University of Bern (Other); Wageningen University (Other); Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Miriam Clegg, Associate Professor, University of Reading
Other Study IDs: UREC 22/29
Record Dates: First submitted 2022-12-15; First posted 2023-01-04 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Older Adults; Appetitive Behaviour; Food Intake; Oral Processing
Keywords: older adults; appetite; oral processing; food intake; chewing; salivary flow; gastric emptying

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about changes in oral processing and appetite in older adults aged 65+ years old. The main question it aims to answer is if oral processing affects gastric emptying in older adults (≥65 years old).

DETAILED DESCRIPTION:
* To investigate if food intake and satiety differ between faster and slower eaters, within older adults (≥65 years old).
* To assess if chewing rate, salivary flow rate, oral processing and gastric emptying differ between older adults (≥65 years old) with smaller versus bigger appetites.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or over (no upper age limit);each group will contain an equal number of male and female participants;
* living sufficiently local to attend the two visits needed;
* able to understand and communicate in English language.

Exclusion Criteria:

* Diagnosed dysphagia;
* (recent) oral surgery that significantly affects eating and/or swallowing;
* diagnosis of type 1 or type 2 diabetes;
* participant undergoing current treatment for cancer;
* participants with zero natural teeth;
* severe loss of appetite and not able to finish a meal (based on CNAQ) and/or people on special or therapeutic diets that restrict the consumption of a full meal and/or the meals provided;
* not able to provide informed consent as defined by the T-CogS test (participants with T-CogS < 22 will be excluded);
* participants having a pacemaker;
* not able to accept the two meal dishes provided and/or relevant food/ingredient included in the meals allergies or intolerances or aversions;
* not able to feed themselves.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy adults aged 65 years old or older
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Objective appetite assessment: Ad-libitum meal consumption | During the procedure
  Consumption of the ad-libitum meal is measured (g). Participants are instructed to eat until they feel comfortable full

SECONDARY OUTCOMES:
Subjective appetite assessment: VAS | During the procedure
  Appetite are assessed using a 100 mm Visual Analogue Scales (VAS, scale 0-100)
Gastric Emptying | During the procedure
  Gastric emptying is measured using of 100 microliters of 13C Octanoic Acid breath test
Chewing rate | During the procedure
  Chewing rate would be assessed with recording the preload breakfast meal provided and analysing the video recording in software (ELAN 6.4) for number of chews, bites, swallows, time of food in the mouth.
Salivary flow rate | During the procedure
  Stimulated and unstimulated salivary flow rate would be assessed with passive drooling method.
BMI | During the procedure
  BMI is assessed by using a body composition monitor (OMRON Viva)
Oral Health | During the procedure
  Oral Health will be assessed by using an Oral Health Questionnaire
Chewing ability | During the procedure
  Chewing ability will be assessed by using a colour mixing ability chewing gum test (Heu-Check test, University of Bern)
Glucose | During the procedure. Every 15 minutes for the first hour after the meal and every 30 minutes thereafter till the end of the total 3 hours
  Glucose will be assessed from finger prick blood samples
Insulin | During the procedure. Every 15 minutes for the first hour after the meal and every 30 minutes thereafter till the end of the total 3 hours
  Insulin will be assessed from finger prick blood samples
Salivary a-amylase | During the procedure
  Salivary a-amylase activity will be assessed from the stimulated saliva collected, by using a-amylase kinetic kit

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Clegg, BSc, PhD, Principal Investigator — m.e.clegg@reading.ac.uk
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however, it is possible that some of the individual (unlinked / non-identifiable) data will be useful in a meta-analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Tada A, Miura H. Systematic review of the association of mastication with food and nutrient intake in the independent elderly. Arch Gerontol Geriatr. 2014 Nov-Dec;59(3):497-505. doi: 10.1016/j.archger.2014.08.005. Epub 2014 Aug 17. PMID 25179444
- [Background] Pina GMS, Mota Carvalho R, Silva BSF, Almeida FT. Prevalence of hyposalivation in older people: A systematic review and meta-analysis. Gerodontology. 2020 Dec;37(4):317-331. doi: 10.1111/ger.12497. Epub 2020 Sep 23. PMID 32965067
- [Background] Morley JE, Silver AJ. Anorexia in the elderly. Neurobiol Aging. 1988 Jan-Feb;9(1):9-16. doi: 10.1016/s0197-4580(88)80004-6. PMID 2898107
- [Background] Krop EM, Hetherington MM, Nekitsing C, Miquel S, Postelnicu L, Sarkar A. Influence of oral processing on appetite and food intake - A systematic review and meta-analysis. Appetite. 2018 Jun 1;125:253-269. doi: 10.1016/j.appet.2018.01.018. Epub 2018 Feb 22. PMID 29408331